CLINICAL TRIAL: NCT05379062
Title: Singing in a Group Compared to Receptive Music and Treatment as a Usual Condition in Patients With Parkinson's Disease: A Randomized Controlled Trial to Develop Guidelines/Recommendations for Efficient Use
Brief Title: Choral Singing for Patients With Parkinson's
Acronym: CHORMORPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salzburg (Other)
Collaborators: University of Vienna (Other); Confraternität Private Hospital (Unknown)
Responsible Party: Principal Investigator, Katarzyna Grebosz-Haring, Principal Investigator, University of Salzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1_1: 2020-06-08
Record Dates: First submitted 2022-04-25; First posted 2022-05-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Parkinson
Keywords: Parkinson; Singing; Music; Stress; Cortisol; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Experimental group (singing in a group/active) Experimental group (receptive music/auditive) Control group (treatment as usual condition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Singing Group (Experimental): Active singing in a group
  Interventions: Behavioral: Active Singing Group
- Receptive Music Group (Experimental): Receptive music/auditive group
  Interventions: Behavioral: Receptive Music Group
- Control Group (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Active Singing Group — The participants of the Active Singing Group take part in a weekly 45-minute singing activity in a group over a period of 3 months. In total the investigators expect 12 choir rehearsals. The rehearsals will take place between 2pm and 3.30pm in the church of the Wehrle-Diakonissen Private Clinic in Salzburg. The group will be led by a professional and experienced choir director.
  Arms: Active Singing Group
Behavioral: Receptive Music Group — The participants of the Receptive Music Group will individually listen to the already researched CD for Parkinson's patients (Bernatzky, Wendtner, Volc, 2012) at home at the same time on one weekday.
  Arms: Receptive Music Group

SUMMARY:
Study Design: Multi-centered, open, prospective, three-arm, randomized, controlled parallel-group study;

Study Participants: Adult patients with Parkinson's disease in Salzburg (and surroundings) and Vienna (and surroundings);

Planned Sample Size: Experimental Group 1 (singing in a group/active): 30 persons; Experimental group 2 (receptive music/auditive): 30 persons; Control group (treatment as usual condition): 30 persons;

Planned Duration of Study: Recruitment: spring 2022, study duration: spring 2022 to autumn 2022, evaluation phase and publication: autumn-summer 2022/2023;

Primary Objectives: Reduction of depression, anxiety and physiological stress; Measurement of the Endpoints: Hospital Anxiety and Depression Scale - German Version (HADS-D), Biochemical determination: cortisol and alpha-amylase (concentration measurement in saliva).

DETAILED DESCRIPTION:
Parkinson's disease is predominantly a disease of old age. A total of about 16,000 patients suffer from Parkinson's disease in Austria. This corresponds to about 0.1% of the population over 50 years of age. In addition to motor and language deficits, psychological deficits also occur. These are usually found between the ages of 50 and 60. The lack of dopamine is the main basis of modern Parkinson therapy. The physiological part of Parkinson's disease can today be well-controlled with medication. Significantly better results can only be achieved with accompanying music-related interventions. For example, regular group singing under professional guidance seems advantageous. The music-induced, rhythmic movement associated with singing, the active posture, the more differentiated strain on the vocal apparatus and breathing compared to speaking, and last but not least, the predominantly positive affectivity show that singing is a complex, ecologically valid form of interpersonal interaction that is also effective on a psychosocial level. In short, many of the therapeutic goals relevant to people with Parkinson's disease are likely to be better achieved through this group activity. Singing together stimulates numerous physical systems as well as perception, attention and cognition. Synchronised movements have also been associated in various studies with increased pain tolerance and may be beneficial in maintaining motor performance in people with Parkinson's disease. Singing improves the immune defence of many patients according to further systematic observations. The results show clear improvements in various health indicators, also in a sustainable course. In addition, regular listening to specifically selected stimulating music, as compiled on a new CD (ISBN: 978-3-9502441-2-0) produced by the project submitter's research group, leads to increased blood flow to certain brain areas. Among other things, dopamine is released. In case of sudden blockages, the pointed rhythm of the Radetzky March, recorded on the CD, helps in a rapid way that could not be achieved with any medication in such a short time.

The aim of this randomized study is to investigate the effect of group singing on the improvement of symptoms of Parkinson's disease, depression, anxiety and stress. Furthermore, the quality of life and the course of parkinson's disease will be assessed. It must also be clarified how often choral singing can be rehearsed in a meaningful way before a weakening (tolerance) of the effect occurs and how high the patients' compliance is. To objectify this study, three groups will be randomly assigned: group one receives the group singing intervention, group two the music listening intervention and group three as a control group (treatment as usual group) receives no musical activity.

The results of the present study should be offered to the rehabilitation centres for support of Parkinson patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Parkinson's disease 1-4 according to Hoehn-Yahr Scale
* Signed consent to participate in the study
* Age >18

Exclusion Criteria:

* Morbus Parkinson 5 according to Hoehn-Yahr Scale
* Dementia
* Aversion to music (Amusia)
* Participation in other active music-based activities (e.g. choir singing, dancing, playing an instrument, making music, playing in an orchestra) during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Anxiety and Depression at 6 and 12 weeks | 18 weeks; outcomes will be measured at the beginning of the study, after 6 weeks, at the end of the study after 12 weeks, and at a follow-up 6 weeks after the end of the study
  Hospital Anxiety and Depression Scale - German Version 2011, C. Herrmann-Lingen, U. Buss & R. P. Snaith. Minimum value 0, maximum value 21, higher score means a better outcome
Change Short-Term Neuroendocrine Stress (Hypothalamic-Pituitary-Adrenal Axis) from pre- to post music interventions over 12 weeks | 12 weeks; outcomes will be measured weekly immediately before and after each 45-minute session in the experimental groups. Outcomes in the control group will be measured twice every week at the same times, 45 minutes apart
  Biological Stress Marker: Salivary Cortisol
Change Short-Term Neuroendocrine Stress (Autonomic Nervous System) from pre- to post music interventions over 12 weeks | 12 weeks; outcomes will be measured weekly immediately before and after each 45-minute session in the experimental groups. Outcomes in the control group will be measured twice every week at the same times, 45 minutes apart
  Biological Stress Marker: Salivary Alpha-Amylase

SECONDARY OUTCOMES:
Mood | 12 weeks; outcomes will be measured weekly immediately before and after each 45-minute session in the experimental groups. Outcomes in the control group will be measured twice every week at the same times, 45 minutes apart
  Multidimensional Mood State Questionnaire, short version (1997), R. Steyer, P. Notz, P. Schwenkmezger & M. Eid. Higher score means a better outcome
Stress Perception | 12 weeks; outcomes will be measured weekly immediately before and after each 45-minute session in the experimental groups. Outcomes in the control group will be measured twice every week at the same times, 45 minutes apart
  Visual Analogue Scale. Minimum 0, Maximum 100, higher score means a worse outcome
Chronic Stress | 18 weeks; outcomes will be measured at the beginning of the study, after 6 weeks, at the end of the study after 12 weeks, and at a follow-up 6 weeks after the end of the study
  Perceived Stress Scale German version (2020), E.E. Schneider, S. Schönfelder, M. Domke-Wolf & M. Wessa. Higher score means a worse outcome
Participation in meetings (compliance) | 12 weeks; outcomes will be measured weekly pre singing intervention
  Self-developed compliance sheet for patients. Minimum 0, maximum 12. Higher score means a better outcome
Life Quality | 18 weeks; outcomes will be measured at the beginning of the study, after 6 weeks, at the end of the study after 12 weeks, and at a follow-up 6 weeks after the end of the study
  Parkinson's Disease Questionnaire German Version (2011), S. Schädler. Minimum 0, maximum 100, higher score means a worse outcome
Consumption of medication | 18 weeks; outcomes will be measured at the beginning of the study, after 6 weeks, at the end of the study after 12 weeks, and at a follow-up 6 weeks after the end of the study
  Sheet for patients, higher score means a worse outcome
Parkinson development | 12 weeks; outcomes will be measured at the beginning of the study and at the end of the study after 12 weeks
  Hoehn-Yahr scale (1967), M. M. Hoehn & M. D. Yahr (evaluation by the neurologist). Minimum value 1, maximum value 5, higher score means a worse outcome
Evaluation of the intervention | 12 weeks; outcomes will be measured weekly post singing and music listening sessions
  Liking of the session, liking of the songs/music pieces, familiarity with the songs/music pieces (9-point Likert scale; higher score means a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Grebosz-Haring, Dr., Principal Investigator — Focus Area Science and Art
Locations (2):
- Austria (2):
  - University of Salzburg / University Mozarteum Salzburg, Salzburg
  - University of Salzburg, Salzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Likar R, Bernatzky G. [Improvement of pain therapy in Austria]. Schmerz. 2007 Jun;21(3):277. doi: 10.1007/s00482-007-0555-2. No abstract available. German. PMID 17632876
- [Result] Bernatzky G, Bernatzky P, Hesse HP, Staffen W, Ladurner G. Stimulating music increases motor coordination in patients afflicted with Morbus Parkinson. Neurosci Lett. 2004 May 6;361(1-3):4-8. doi: 10.1016/j.neulet.2003.12.022. PMID 15135879
- [Result] Grebosz-Haring K, Schuchter-Wiegand AK, Feneberg AC, Skoluda N, Nater UM, Schutz S, Thun-Hohenstein L. The Psychological and Biological Impact of "In-Person" vs. "Virtual" Choir Singing in Children and Adolescents: A Pilot Study Before and After the Acute Phase of the COVID-19 Outbreak in Austria. Front Psychol. 2022 Jan 4;12:773227. doi: 10.3389/fpsyg.2021.773227. eCollection 2021. PMID 35058843
- [Result] Grebosz-Haring K, Thun-Hohenstein L. Effects of group singing versus group music listening on hospitalized children and adolescents with mental disorders: A pilot study. Heliyon. 2018 Dec 17;4(12):e01014. doi: 10.1016/j.heliyon.2018.e01014. eCollection 2018 Dec. PMID 30582039
- [Result] Grebosz-Haring K, Thun-Hohenstein L, Schuchter-Wiegand AK, Irons Y, Bathke A, Phillips K, Clift S. The Need for Robust Critique of Arts and Health Research: Young People, Art Therapy and Mental Health. Front Psychol. 2022 Feb 10;13:821093. doi: 10.3389/fpsyg.2022.821093. eCollection 2022. PMID 35222203
- [Result] Panksepp J, Bernatzky G. Emotional sounds and the brain: the neuro-affective foundations of musical appreciation. Behav Processes. 2002 Nov;60(2):133-155. doi: 10.1016/s0376-6357(02)00080-3. PMID 12426066